CLINICAL TRIAL: NCT06371131
Title: Effect of Right⁃Stellate Ganglion Block on Postoperative Nausea and Vomiting in Patients Undergoing Thyroid Surgery
Brief Title: Effect of Stellate Ganglion Block on Postoperative Nausea and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: PONV of Thyroid Surgery
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-04

CONDITIONS: Stellate Ganglion Block; Thyroid Surgery; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Experimental group: right stellate ganglion block 30 minutes before anesthesia induction.Control group: No treatment was given 30minutes before anesthesia induction.Data was recorded at the corresponding time points.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right stellate ganglion block (Experimental): Right -stellate ganglion block was given 30minutes before anesthesia induction.
  Interventions: Procedure: Right -stellate ganglion block
- Blank control group (No Intervention): No treatment was given 30 minutes before anesthesia induction

INTERVENTIONS:
Procedure: Right -stellate ganglion block — The experimental group was given right stellate ganglion block 30 minutes before anesthesia induction
  Arms: Right stellate ganglion block

SUMMARY:
Postoperative nausea and vomiting is one of the most common postoperative complications second only to postoperative pain. Studies have reported that without any antiemetic prevention treatment, the overall incidence of PONV in surgical operations is up to 20-30%, and the incidence of PONV in high-risk patients such as thyroid surgery is even up to 70-80%. PONV not only increased discomfort and prolonged hospital stay; Severe cases can lead to wound dehysis, acid-base imbalance, water and electrolyte metabolism disorders, seriously affect the prognosis of patients. Although various prevention and treatment measures have been adopted in clinical practice, it still cannot be completely eliminated. Therefore, postoperative nausea and vomiting of thyroid is still a concern in clinical anesthesia work, so it is urgent to explore more simple and effective measures to prevent thyroid PONV. SGB is the injection of local anesthetics into loose connective tissue containing stellate ganglion. It has a clear effect on postoperative analgesia of thyroid surgery, and can play a certain role in preventing thyroid PONV by reducing the application of perioperative opioids. Few studies have reported that the incidence of PONV can be significantly reduced after the application of SGB in patients with thyroid surgery, which provides a certain basis for the prevention of thyroid PONV. Therefore, this study aims to explore the effect of right stellate ganglion block on preventing postoperative nausea and vomiting of thyroid, and to explore the possible mechanism of action.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting is one of the most common postoperative complications second only to postoperative pain. Studies have reported that without any antiemetic prevention treatment, the overall incidence of PONV in surgical operations is up to 20-30%, and the incidence of PONV in high-risk patients such as thyroid surgery is even up to 70-80%. The pathogenesis of postoperative nausea and vomiting is very complex, including central, peripheral receptors and multiple nerve pathways. When peripheral receptors are stimulated, the signal passes through the afferent nerve to the vomiting center, causing nausea and vomiting. The emetic chemical receptors are rich in many receptors, which can directly feel various toxins, metabolites or drugs in the blood and cerebrospinal fluid, project signals to the nerve center and then spread to the cerebral cortex, causing nausea and vertigo, or transmit signals along the vagus nerve, glossopharyngeal nerve, spinal nerve, etc. to the digestive tract, diaphragm and abdominal wall muscles, resulting in the opening of the sphincter in the upper esophagus and strong contraction of the diaphragm. Abdominal muscles contract, so that the stomach pressure increases, stomach contents through the digestive tract is expelled from the body, vomiting.

Thyroid, as the endocrine organ of human body, mainly secretes thyroid hormone and participates in human metabolism. With the progress of modern medical technology, although thyroid postoperative complications have decreased, due to the limited operating space of thyroid surgery, in order to fully exposed the surgical field of vision and facilitate the operation of surgeons, patients often take the cervical hyperextension position, that is, patients take the supine position with high shoulder pads. Tilt your head back so that your lower jaw, trachea, and sternum are at the same level, allowing the thyroid gland to protrate forward as much as possible. Although this position is easy for surgeons to operate, due to the complex anatomical structure around the thyroid gland, adjacent to important blood vessels and nerves, this position often causes thyroid surgical position syndrome in patients, that is, nausea and vomiting, dizziness, headache, tinnitus, neck radiation pain and other symptoms, which not only increases patients' pain, but also seriously reduces patients' medical experience.

Stellate ganglion block has been proved to be widely used in clinic and can play a positive role in multiple organs and systems of the whole body. In clinical work, stellate ganglion block is more widely used in the treatment of various pain, autonomic nerve disorders and other diseases. However, there are few clinical studies on whether stellate ganglion block can be used as an effective and feasible means to prevent postoperative nausea and vomiting and the related mechanisms to prevent the possible occurrence of nausea and vomiting. Therefore, this study will explore the preventive effect of stellate ganglion block on postoperative thyroid nausea and vomiting, and hope to explore its possible mechanism, so as to provide more effective and feasible methods for clinical prevention of postoperative nausea and vomiting and improve patients' medical comfort and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving thyroid surgery under general anesthesia
2. Age ≥18 years and ≤ 70 years
3. American Society of Anesthesiologists(ASA) physical status classification I-III.
4. Voluntary participation and ability to understand and sign the informed consent form.

Exclusion Criteria:

1. Patients with obesity(BMI>30 kg/m2)
2. contraindicated to stellate ganglion block
3. Patients who cannot cooperate with the study for any reason, or whom the investigator deems unsuitable for inclusion in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative nausea and vomiting | From end of surgery to 24 hours after surgery
  Postoperative nausea and vomiting is evaluated by follow-up

SECONDARY OUTCOMES:
Incidence of Postoperative nausea and vomiting during preemptive analgesia | From 0-10 min after preemptive analgesia
  Postoperative nausea and vomiting is evaluated by investigator's follow-up
Intensity of nausea and vomiting during preemptive analgesia | From 0-10 min after preemptive analgesia
  Intensity of nausea and vomiting is evaluated by numeric rating scale (0-10), which higher socre represents more uncomfortable
Intensity of nausea and vomiting during hospitalization | From end of surgery to 24 hours after surgery
  Intensity of nausea and vomiting is evaluated by numeric rating scale (0-10), which higher socre represents more uncomfortable
Hemodynamic parameters after preemptive analgesia | From 0-10 min after preemptive analgesia
  Systolic blood pressure，dastolic blood pressure，mean arterial pressure，heart rate，oxygen saturation，Patient state index
Postoperative pain intensity | From end of surgery to 24 hours after surgery
  Postoperative pain intensity is assessed by numeric rating scale (0-10), which higher socre represents more uncomfortable
Recovery of gastrointestinal function | From end of surgery to 24 hours after surgery
  Gastrointestinal function is is assessed by the evacuation time
Sleep quality | From end of surgery to 1 day after surgery
  Sleep quality is is assessed by numeric rating scale (0-10), which higher socre represents better sleep quality
Satisfaction score and postoperative analgesia satisfaction score | From end of surgery to hospital discharge with about 5 days
  Satisfaction score and postoperative analgesia satisfaction score is assessed by numeric rating scale (0-10), which higher socre represents more uncomfortable

CONTACTS AND LOCATIONS:
Overall Officials: ling Dan, BD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication